CLINICAL TRIAL: NCT06639802
Title: Effects of Hand Arm Bimanual Intensive Therapy Including Lower Extremity on Balance and Coordination in Ataxic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/31
Record Dates: First submitted 2024-09-20; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ataxic Cerebral Palsy; Coordination and Balance Disturbances
Keywords: Physical Therapy Technique; coordination impairement; Ataxic Cerebral Palsy; HAnd Arm Bimanual Intensive Therapy including Lower Extremity
MeSH Terms: conditions — Cerebral Palsy, Ataxic, Autosomal Recessive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): HABIT-ILE is continuous intervention applied for 50-90 hours over two weeks. We will design the activities based on the findings of the initial assessments (T0) T0he customized functional goals that were previously discussed with the parents (e.g., drinking on one's own without spilling, using one hand to hold a book while turning pages with the other, removing a t-shirt, etc.).
  The whole environment is arranged in such a way that children perceive the therapy as fun.
  Progression of difficulty depend upon success in performance of current level. Specific bi-manual activities are selected on basis of child's motor abilities, age and interest.
  Interventions: Other: Hand Arm Bimanual Intensive therapy including lower extremity (HABIT-ILE)

INTERVENTIONS:
Other: Hand Arm Bimanual Intensive therapy including lower extremity (HABIT-ILE) — HABIT-ILE is continuous intervention applied for 50-90 hours over two weeks. We will design the activities based on the findings of the initial assessments (T0) and the customized functional goals that were previously discussed with the parents (e.g., drinking on one's own without spilling, using one hand to hold a book while turning pages with the other, removing a t-shirt, etc.). HABIT-ILE activities are presented as games and the whole environment is arranged in such a way that children perceive the therapy as fun. Progression of difficulty depend upon success in performance of current level. Specific bi-manual activities are selected on basis of child's motor abilities, age and interest.

SUMMARY:
Ataxic cerebral palsy is an abnormal movement or posture pattern accompanied by a loss of coordinated muscle action, resulting in movements that lack proper force, rhythm, or accuracy. Ataxic CP is classified into cerebellar ataxia and ataxic diplegia.

In Cerebellar Ataxia, the cerebellum is hypo-plastic or malformed which impairs the integration of brain signals required for coordinating coordinated movement and balance. This study aimed to determine the effect of HABIT-ILE on the balance and coordination of children with cerebellar ataxic cerebral palsy.

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To determine the effect of HABIT-ILE on the coordination of children with cerebellar ataxic cerebral palsy.
2. To determine the effect of HABIT-ILE on the balance of children with cerebellar ataxic cerebral palsy.

HYPOTHESIS:

Alternate Hypothesis:

There will be statistically significant differences in balance and coordination after HABIT-ILE in ataxic cerebral palsy.(P>0.05)

Null Hypothesis:

There will be no statistically significant differences in balance and cooordination after HABIT-ILE in ataxic cerebral palsy.(P>0.05)

Research Design: Experimental study. Quasi-experimental

Clinical setting: Al-Farabi Special Education Institute Islamabad Study duration: one year from Feb 2024 to 2025.

Selection Criteria:

Inclusion Criteria

1. Age group: 6 - 15 years.
2. Gender: Both males and females.
3. Cerebellar Ataxic cerebral palsy [1]
4. Gross motor function classification system level I and II.
5. Capable of following instructions and completing all necessary tests and tasks

Exclusion Criteria

1. Uncontrolled epilepsy
2. Orthopedic surgery within the past 6 months,
3. Have visual, hearing impairments (diagnosed).

Sampling technique: convenicence sampling

Outcome Measures:

1. Pediatric Balance Scale [2]
2. Scale for the Assessment and Rating of Ataxia [3]
3. Gross Motor Function Classification System - Expanded & Revised (GMFCS - E&R) [4]

Data analysis techniques:

Data will be analyzed using SPSS version 20.0.0.

Significance of the study:

Cerebellar ataxic cerebral palsy is characterized by hypoplasia or malformations of the cerebellum, which hinders the integration of neural information necessary for coordination and balance.

HABIT-ILE aims to collectively target the whole body both upper and lower extremity along with trunk in intensive therapy comprising of fun and playful goal oriented tasks in order to improve balance and coordination.

So this research will find out effects of HABIT-ILE on balance and coordination of children with cerebellar ataxic cerebral palsy. Positive research outcome can contribute to better independence.

This study will add data in the limited literature of ataxic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 6 - 15 years.
* Gender: Both males and females.
* Cerebellar Ataxic cerebral palsy [10]
* Gross motor function classification system level I and II.
* Capable of following instructions and completing all necessary tests and tasks

Exclusion Criteria:

* Uncontrolled epilepsy
* Orthopedic surgery within the past 6 months,
* Have visual, and hearing impairments (diagnosed).

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Balance | 2 weeks
  A modified version of the Berg Balance Scale, the Pediatric Balance Scale is used to evaluate school-age children's functional balance abilities. The 14 items on the scale have a maximum score of 56 points and are rated from 0 (lowest function) to 4 (highest function).
Coordination | 2 weeks
  Method for evaluating ataxia is SARA, which consists of eight categories, each category is scored from 0 (no ataxia) to 40 (severe ataxia) based on the performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No